CLINICAL TRIAL: NCT01644760
Title: Respiratory Variations in the Diameter of the Inferior Vena Cava With Spontaneous Ventilation: A Physiological Study on Healthy Volunteers
Brief Title: Respiratory Variations in the Diameter of the Inferior Vena Cava With Spontaneous Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2012/LM-01; 2012-A00625-38 (Other: ANSM)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-03

CONDITIONS: Collapsibility of the Inferior Vena Cava
Keywords: Diaphragmatic excursion; normality
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study population (Experimental): Healthy subjects with spontaneous ventilation, 18 to 50 years of age.
  Interventions: Procedure: Ultrasounds with controlled breathing

INTERVENTIONS:
Procedure: Ultrasounds with controlled breathing — The patient will have cardiac, abdominal and thoracic ultrasounds with controlled and monitored inspiratory effort. This gesture takes about 40 minutes.

SUMMARY:
The main objective of this study is to determine a threshold value of diaphragmatic excursion (ultrasound measures: expiration versus inspiration)that best predicts a 50% collapsibility of the inferior vena cava.

DETAILED DESCRIPTION:
Secondary objectives of this study are:

* to determine a threshold value of diaphragmatic excursion (ultrasound measures: expiration versus inspiration)that best predicts a 40% collapsibility of the inferior vena cava (IVC).
* to determine a threshold value of diaphragmatic excursion (ultrasound measures: expiration versus inspiration)that best predicts a 100% collapsibility of the IVC.
* to determine the location of the cutting plane for the TM analysis of collapsibility of the IVC.
* to evaluate the hemodynamic conditions of normal healthy volunteers.
* to detect any abnormality of cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* The volunteer must have given his/her informed and signed consent
* The volunteer must be insured or beneficiary of a health insurance plan

Exclusion Criteria:

* The volunteer is participating in another study
* The volunteer is in an exclusion period determined by a previous study
* The volunteer is under judicial protection, under tutorship or curatorship
* The volunteer refuses to sign the consent
* It is impossible to correctly inform the volunteer
* The patient is pregnant, parturient, or breastfeeding
* The volunteer has known heart disease like heart failure, cardiac arrhythmia
* The volunteer takes cardiotropics
* The volunteer has known lung disease: obstructive or restrictive respiratory failure
* The volunteer has clinical signs of COPD (coughing with morning sputum in a smoking subject)
* Any emergency situation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09-17 (Actual); Study Completion 2012-09-17 (Actual)

PRIMARY OUTCOMES:
Collapsibility score for the IVC diameter | Baseline (Day 0; cross-sectional study)
  percentage = ((max-min)/average)*100%
  Three variables are necessary to respond to the primary objective: (the collapsibility score for the IVC diameter; (2) whether or not this score is >= 50%; and (3) a measure of the diaphragmatic excursion.
Collapsibility score for the IVC diameter >= 50% (presence/absence) | Baseline (Day 0; cross-sectional study)
  percentage = ((max-min)/average)*100%
  Three variables are necessary to respond to the primary objective: (the collapsibility score for the IVC diameter; (2) whether or not this score is >= 50%; and (3) a measure of the diaphragmatic excursion.
Diaphragmatic excursion | Baseline (Day 0; cross-sectional study)
  Maximum distance between the position of the diaphragmatic dome during inspiration versus expiration (cm)
  Three variables are necessary to respond to the primary objective: (the collapsibility score for the IVC diameter; (2) whether or not this score is >= 50%; and (3) a measure of the diaphragmatic excursion.

SECONDARY OUTCOMES:
Collapsibility score for the IVC diameter >= 40% (presence/absence) | Baseline (Day 0; cross sectional study)
  percentage = ((max-min)/average)*100%
Collapsibility score for the IVC diameter >= 60% (presence/absence) | Baseline (Day 0; cross sectional study)
  percentage = ((max-min)/average)*100%
Mitral Doppler Wave E speed | Baseline (Day 0; cross sectional study)
  cm/s
Mitral Doppler Wave A speed | Baseline (Day 0; cross sectional study)
  cm/s
Tissue Doppler Wave E' speed | Baseline (Day 0; cross sectional study)
  cm/s
Simpson: FEVG | Baseline (Day 0; cross sectional study)
  %

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Muller, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Gignon L, Roger C, Bastide S, Alonso S, Zieleskiewicz L, Quintard H, Zoric L, Bobbia X, Raux M, Leone M, Lefrant JY, Muller L. Influence of Diaphragmatic Motion on Inferior Vena Cava Diameter Respiratory Variations in Healthy Volunteers. Anesthesiology. 2016 Jun;124(6):1338-46. doi: 10.1097/ALN.0000000000001096. PMID 27003619